CLINICAL TRIAL: NCT06500780
Title: Equipping Patients Using Interventions for Pain and Depression (EQUIPD) - Phase 2
Brief Title: Equipping Patients Using Interventions for Pain and Depression
Acronym: EQUIPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Adam Todd Hirsh, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22412; 4R33NR020845-02 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Depression; Health Equity
Keywords: chronic pain; depression; health equity; shared decision making; decision aid; depressive symptoms
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Depression | interventions — Decision Support Techniques

STUDY DESIGN:
Masking Description: Baseline assessments are conducted prior to randomization (Baseline assessor will not know the randomization assignment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching and Decision Aid (Experimental): Intervention group (Individual coaching sessions and Decision Aid)
  Interventions: Behavioral: Coaching and Decision Aid
- Control (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: Coaching and Decision Aid — Four (4) coaching sessions over approximately 12 weeks with integration of Decision Aid contents
  Arms: Coaching and Decision Aid

SUMMARY:
This project is part of the NIH Helping to End Addiction Long-term (HEAL) initiative (https://heal.nih.gov/). This randomized controlled trial (RCT) is phase 2 of a two-phase, 5-year project with the overarching goal of testing a decision aid (DA)/coaching intervention, tailored to Black patients with comorbid chronic pain and depression, to encourage use of and adherence to nonpharmacological pain treatments (NPTs).

This 2-arm trial will randomize 304 patients with comorbid chronic musculoskeletal pain and depression in primary care from an urban safety-net health system (Eskenazi). After the baseline assessment, patients randomized to the intervention will be asked to participate in 4 coaching sessions over approximately 12 weeks. Sessions will use Motivational Interviewing principles to foster openness to NPTs and self-efficacy by helping patients identify their goals and priorities, understand their NPT options, prepare them to discuss and choose options with their primary care providers (PCPs), and reinforce these choices to foster maintenance of these changes. DA contents will be integrated into these sessions, which will facilitate discussion of these options with their PCP. The first 3 sessions take place prior to the patient's next scheduled PCP visit; the final session occurs after this visit. Assessments will be conducted at baseline, 3 months (i.e., after completing the final coaching session), and 6 months.

Patients randomized to the wait-list control group will receive usual care (in addition to study assessments at baseline, 3 months, and 6 months). After completing the final assessment, they will then be given the DA and offered a 20-minute coaching session to walk them through it.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must

* have musculoskeletal pain in the low back, cervical spine, or extremities (hip, knee, shoulder) for ≥3 months,
* have at least moderate pain intensity and interference with function, defined by a score ≥4 (possible range: 0-10) on the Pain, Enjoyment of Life and General Activity scale (PEG), a 3-item measure of pain intensity, interference with enjoyment of life, and interference with general activity,
* have at least mild depression, defined as PHQ-8 score ≥5,
* identify as Black or African American,
* have consistent access to a telephone,
* indicate openness to new pain treatments, and
* have a scheduled appointment with their PCP in the next approximate 2-4 months or be willing to schedule one

Exclusion Criteria:

Patients are excluded:

* if previously participated in Dr. Matthias' past pilot study (IRB #12885), the pilot RCT for this project (IRB #16571), or are participating as a Patient Engagement Panel member for this project (Aim 1.1),
* if the eligibility screener or medical records indicate severe medical conditions likely precluding participation (e.g. stroke in the last 6 months, hospitalized with congestive heart failure or a heart attack in the last 6 months, cancer other than skin cancer and receiving active treatment), or
* if the eligibility screener or medical records reveal (1) active suicidal ideation, or (2) severe hearing/speech or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Brief Pain Inventory (BPI) Interference Scale at 3 months | 3 months
  The pain interference score averages seven ratings, 0 (does not interfere) to 10 (completely interferes).
Change from Baseline Brief Pain Inventory (BPI) Interference Scale at 6 months | 6 months
  The pain interference score averages seven ratings, 0 (does not interfere) to 10 (completely interferes).
Change from Baseline Patient Health Questionnaire (PHQ)-8 at 3 months | 3 months
  The Patient Health Questionnaire (PHQ)-8 is a widely-used, validated 8-item measure of depression severity that uses a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Change from Baseline Patient Health Questionnaire (PHQ)-8 at 6 months | 6 months
  The Patient Health Questionnaire (PHQ)-8 is a widely-used, validated 8-item measure of depression severity that uses a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).

SECONDARY OUTCOMES:
Change from Baseline Generalized Anxiety Disorder (GAD)-7 at 3 months | 3 months
  Anxiety will be measured with the 7 item Generalized Anxiety Disorder (GAD)-7 that uses a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Change from Baseline Generalized Anxiety Disorder (GAD)-7 at 6 months | 6 months
  Anxiety will be measured with the 7 item Generalized Anxiety Disorder (GAD)-7 that uses a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Change from Baseline Pain Catastrophizing Scale at 3 months | 3 months
  The Pain Catastrophizing Scale is a 13-item scale that assesses catastrophizing-a cognitive-emotional factor that predicts poor treatment response. The scale uses a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time).
Change from Baseline Pain Catastrophizing Scale at 6 months | 6 months
  The Pain Catastrophizing Scale is a 13-item scale that assesses catastrophizing-a cognitive-emotional factor that predicts poor treatment response. The scale uses a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time).
Change from Baseline Use of Nonpharmacological and Self-Care Approaches (NSCAP) at 3 months | 3 months
  The NSCAP asks about 9 nonpharmacological treatment (NPT) modalities and assesses details of use such as frequency, location/source of service, and patients' judgments of effectiveness. Space is also provided for other NPTs that are used but not listed. The number of modalities for which patients answer "yes" will be summed for analyses.
Change from Baseline Use of Nonpharmacological and Self-Care Approaches (NSCAP) at 6 months | 6 months
  The NSCAP asks about 9 nonpharmacological treatment (NPT) modalities and assesses details of use such as frequency, location/source of service, and patients' judgments of effectiveness. Space is also provided for other NPTs that are used but not listed. The number of modalities for which patients answer "yes" will be summed for analyses.
Change from Baseline Altarum Consumer Engagement (ACE) Measure at 3 months | 3 months
  Patient engagement will be measured with the 12-item Altarum Consumer Engagement (ACE) Measure, which has 3 subscales: 1) commitment to manage one's health, 2) informed choice, and 3) confidence to participate in treatment decisions. Items are assessed on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).
Change from Baseline Altarum Consumer Engagement (ACE) Measure at 6 months | 6 months
  Patient engagement will be measured with the 12-item Altarum Consumer Engagement (ACE) Measure, which has 3 subscales: 1) commitment to manage one's health, 2) informed choice, and 3) confidence to participate in treatment decisions. Items are assessed on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).
Change from Baseline Decisional Conflict Scale (DCS) at 3 months | 3 months
  Decisional conflict will be measured with the 16-item Decisional Conflict Scale that measures personal perceptions of a) uncertainty in choosing options, b) modifiable factors contributing to uncertainty, and c) effective decision making on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).
Change from Baseline Decisional Conflict Scale (DCS) at 6 months | 6 months
  Decisional conflict will be measured with the 16-item Decisional Conflict Scale that measures personal perceptions of a) uncertainty in choosing options, b) modifiable factors contributing to uncertainty, and c) effective decision making on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree).

OTHER OUTCOMES:
Change from Baseline Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) at 3 months | 3 months
  Communication self-efficacy will be measured with this 5-item scale that measures patients' self-efficacy in obtaining medical information and getting their most important health concern discussed in a clinic visit. The scale uses ratings from 0 (not at all confident) to 10 (extremely confident).
Change from Baseline Perceived Efficacy in Patient-Physician Interactions Scale (PEPPI-5) at 6 months | 6 months
  Communication self-efficacy will be measured with this 5-item scale that measures patients' self-efficacy in obtaining medical information and getting their most important health concern discussed in a clinic visit. The scale uses ratings from 0 (not at all confident) to 10 (extremely confident).

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hirsh, PhD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health Primary Care, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH intends to maximize the impact of HEAL Initiative-supported projects through broad and rapid data sharing. All HEAL Initiative award recipients, regardless of the amount of direct costs requested for any one year, are required to comply with the HEAL Public Access and Data Sharing Policy, which also aligns with the NIH Policy for Data Management and Sharing (https://grants.nih.gov/grants/guide/notice-files/NOT-OD-21-013.html). HEAL award recipients must following all requirements and timelines developed through the HEAL Initiative Data Ecosystem, as described in HEAL's compliance guidance (https://heal.nih.gov/data/complying-heal-data-sharing-policy).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication of the primary manuscript
Access Criteria: Implementation of the plan will follow the HEAL Public Access and Data Sharing Policy.
URL: https://heal.nih.gov/data/public-access-data